CLINICAL TRIAL: NCT02483546
Title: High Fidelity Simulation In Medecine Education
Brief Title: High Fidelity Simulation vs Standard Teaching Training of Cardiac Resuscitation
Acronym: SIMCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 12345
Record Dates: First submitted 2015-02-20; First posted 2015-06-29 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Cardiac Arrest
Keywords: Medical education; simulation; ACLS
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- huma patient based training (Experimental): Students randomized to receive simulation training .The mannequin Siman 3G laerdal® displays multiple physiologic and pharmacologic responses. Three volunteers were involved in the scenario while the others were observers through an audiovisual projection. Students participating in the scenario were given 15 minutes to evaluate and manage a 60-year-old man with a known history of coronary artery disease and diabetes who presented to the emergency department with chest pain revealing an acute ST elevation myocardial infarction complicated by ventricular fibrillation. Students were required to recognize and manage ventricular fibrillation when the patient became pulseless and unresponsive. After performing the simulation, the entire group was convened for debriefing of the case.
  Interventions: Device: Laerdal®; Behavioral: huma patient based training
- traditionally teaching (Active Comparator): students received a traditional course using slides during 60 minutes about the management of cardio pulmonary resuscitation according to the latest recommendations of the AHA. This course is offered by the same trainer who participated in the simulation session. Students were free to ask questions as the progress of education. The same educational objectives were treated with the two groups.
  Interventions: Behavioral: traditionally teaching

INTERVENTIONS:
Device: Laerdal® — simulation- based educational intervention
  Arms: huma patient based training
Behavioral: huma patient based training — Students randomized to receive simulation training .The mannequin Siman 3G laerdal® displays multiple physiologic and pharmacologic responses. Three volunteers were involved in the scenario while the others were observers through an audiovisual projection. Students participating in the scenario were given 15 minutes to evaluate and manage a 60-year-old man with a known history of coronary artery disease and diabetes who presented to the emergency department with chest pain revealing an acute ST elevation myocardial infarction complicated by ventricular fibrillation. Students were required to recognize and manage ventricular fibrillation when the patient became pulseless and unresponsive. After performing the simulation, the entire group was convened for debriefing of the case.
  Arms: huma patient based training
Behavioral: traditionally teaching — Control group students received a traditional course using slides during 60 minutes about the management of cardio pulmonary resuscitation according to the latest recommendations of the AHA. This course is offered by the same trainer who participated in the simulation session. Students were free to ask questions as the progress of education. The same educational objectives were treated with the two groups.
  Arms: traditionally teaching

SUMMARY:
High fidelity Simulation has spread from anesthesiology to other disciplines such as internal medicine, pediatrics, and emergency medicine . Over the past decade, the use of simulation in medical education has increased exponentially. The term ''simulation'' spans a wide variety of formats, from the low-tech actor portraying a standardized patient to high-fidelity mannequin-based human patient simulation (HPS). HPS is able of both simulating realistic patient encounters and giving real-time, physiologically accurate feedback. Studies thus far show that use of simulation in training medical students and residents is helpful in strengthening students' knowledge and in evaluating their performance. Students appreciate simulation-based education as ''an opportunity to learn new skills in a safe environment .

DETAILED DESCRIPTION:
This was a randomized, controlled trial of a simulation- based educational intervention designed to increase medicine student's clinical skills in cardiac arrest procedures .The investigators included 181 fifth-year medical students rotating in the emergency department of Fattouma Bourguiba University hospital of Monastir (Tunisia) during the period from January 2013 to January 2014.Students were randomized into two groups using a random number generator to an intervention group (simulatortrained, n = 99) or a control group (traditionally teaching, n =82).

The investigators conducted a prospective, randomized, non-blinded study to determine whether simulation based training is superior to traditional teaching in the assessment and management of simulated patients presenting with myocardial infarction (MI) complicated by ventricular fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Medecine students

Exclusion Criteria:

* Non Medecine students

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
better acquisition of cognitive skills for students | just after randomisation (one day)
  Pretest using 20 multiple choice questions after randomization. A second round of the same testing was then conducted for both groups just after the course (posttest). The test score range from 0 to 20 (maximum). The difference between the rating of the post-test and pre-test identifies the delta score of the student.

SECONDARY OUTCOMES:
Satisfaction 5 point likert scale | just after randomisation (one day)
  Students rated their satisfaction level with a 5 point likert scale framed as attitude toward simulation compared with control group: dissatisfied (1 point), fairly satisfied (2 points), neither satisfied (3points), satisfied (4 points), and very satisfied (5 points).

CONTACTS AND LOCATIONS:
Overall Officials: Hamdi Boubaker, MD, Principal Investigator — Emergency Department , university Hospital of Monastir 5000 TUNISIA; Mohamed habib GRISSA, MD, Principal Investigator — Emergency Department , university Hospital of Monastir 5000 TUNISIA
Locations (1):
- university of Monastir, Monastir, Monastir Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided